CLINICAL TRIAL: NCT05669976
Title: Suicide Prevention for Sexual and Gender Minority Youth (Randomized Controlled Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Blashill, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-2022-0204; R33MH120236 (NIH)
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Suicide
Keywords: Sexual and gender minority youth; Prevention; Patient Navigation; Safety Planning Intervention
MeSH Terms: conditions — Suicide; Coitus

STUDY DESIGN:
Intervention Model Description: Prospective participants will be recruited within Southern California and requested to fill out a brief online survey. A trained member of the study team will contact each potential participant to explain the study, obtain verbal consent for pre-enrollment screening, and conduct the screening process. For those who meet screening criteria, a trained member of the study team will provide more information about the study and engage in an informed consent process during a virtual appointment. Following informed consent, participants will complete self-report questionnaires and clinician-based interviews. When eligible, participants will be randomized to either receive the PN+SPI intervention or SPI alone and offered virtual appointments. At baseline, 3-month, 6-month, and 12-month follow-ups, participants will complete clinical interviews to assess for suicidal ideation and suicidal behaviors and complete measures of suicidal coping and thwarted belongingness.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors (for primary endpoint: suicide attempts) will be masked for randomized study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Planning Intervention with Navigation Services (Experimental): A patient navigation (PN) intervention for SGM youth/emerging adults designed to target mechanisms (i.e., decreasing thwarted belongingness and increasing suicide-related coping skills) that theoretically underlie suicide. The proposed intervention integrates a single-session, empirically supported, suicide prevention intervention (Safety Planning Intervention; SPI) with PN services (PN+SPI). The patient navigator will deliver the SPI and continue frequent contact for the purpose of providing motivational enhancement, problem-solving, reinforcing coping strategies, and connecting participants to mental health and social support resources (e.g., SGM-specific support groups within the community).
  Interventions: Behavioral: Safety Planning Intervention with Navigation Services
- Safety Planning Intervention (Active Comparator): The Safety Planning Intervention (SPI) is a single-session, empirically supported, suicide prevention intervention. The patient navigator will deliver the SPI.
  Interventions: Behavioral: Safety Planning Intervention

INTERVENTIONS:
Behavioral: Safety Planning Intervention with Navigation Services — A patient navigation (PN) intervention for SGM youth/emerging adults designed to target mechanisms (i.e., decreasing thwarted belongingness and increasing suicide-related coping skills) that theoretically underlie suicide. The proposed intervention integrates a single-session, empirically supported, suicide prevention intervention (Safety Planning Intervention; SPI) with PN services (PN+SPI). The patient navigator will deliver the SPI and continue frequent contact for the purpose of providing motivational enhancement, problem-solving, reinforcing coping strategies, and connecting participants to mental health and social support resources (e.g., SGM-specific support groups within the community).
  Other Names: PN+SPI
  Arms: Safety Planning Intervention with Navigation Services
Behavioral: Safety Planning Intervention — The Safety Planning Intervention (SPI) is a single-session, empirically supported, suicide prevention intervention. The patient navigator will deliver the SPI.
  Other Names: SPI
  Arms: Safety Planning Intervention

SUMMARY:
The overarching goal of this study is to evaluate a newly-developed suicide prevention program for sexual and gender minority youth and emerging adults. After development of the intervention program, a randomized controlled trial will be conducted to test its preliminary efficacy in lowering the risk for suicide attempts.

DETAILED DESCRIPTION:
Suicide is the 10th leading cause of death among all U.S. citizens, and is the 2nd leading cause of death among youth and emerging adults between the ages of 15 and 34. Moreover, U.S. representative data indicate increasing trends in suicide attempts and death by suicide. In addition to the immense psychological burden experienced by the family and friends of individuals who attempt and complete suicide, the costs of death by suicide and suicide attempts in 2013 were estimated at $93.5 billion.

One group that is particularly vulnerable to suicide is sexual and gender minorities (SGMs). SGM is an umbrella term used to describe individuals who identify as non-exclusively heterosexual (e.g., gay, lesbian, bisexual) and/or as transgender/non-binary (e.g., identify as a gender different from their birth sex). Extant research consistently notes substantial mental health disparities among SGMs in comparison to their heterosexual and cis-gender counterparts. In 2017, in the U.S., 23% of sexual minority youth reported one or more suicide attempts (in the past 12 months) vs. 5.4% of heterosexual youth. This disparity has also been noted in a meta-analysis of population-based longitudinal studies, with sexual minority adolescents and emerging adults reporting 2.26 increased odds of suicide attempts compared to their heterosexual counterparts. Prevalence of lifetime suicide attempts among gender minorities is also substantially elevated compared to the general population, with 45% of 18-24-year-old transgender individuals reporting history of one or more suicide attempts.

Despite these substantial health disparities in suicide among SGM youth/emerging adults, no known suicide prevention programs exist for this highly vulnerable population. Given this crucial gap in the literature, the proposed study will adapt and test a patient navigation (PN) intervention for SGM youth/emerging adults designed to target mechanisms (i.e., decreasing thwarted belongingness and increasing suicide-related coping skills) that theoretically underlie suicide. The intervention integrates a single-session, empirically supported, suicide prevention intervention (Safety Planning Intervention; SPI) with PN services (PN+SPI). The patient navigator will deliver the SPI and continue frequent contact for the purpose of providing motivational enhancement, problem-solving, reinforcing coping strategies, and connecting participants to social support and mental health resources (e.g., SGM-specific support groups within the community). After completing the development of the PN+SPI intervention during a previous phase of the project, this study will accomplish the following specific aims:

Specific Aim 2: To conduct a pilot randomized controlled trial of the integrated PN+SPI by comparing it to the safety planning intervention alone to assess feasibility, acceptability, and preliminary efficacy. We plan to randomize 170 SGM youth/emerging adults to either the PN+SPI or SPI alone and follow participants for 12 months. It is expected that the pilot trial will provide additional information about the feasibility and acceptability of the PN+SPI intervention and study methods, in preparation for a future full-scale efficacy trial. In addition, the pilot test will evaluate its preliminary impact on suicide attempts. It is hypothesized that participants assigned to the PN+SPI intervention will demonstrate lower suicide attempts in comparison to participants assigned to the SPI alone condition.

Specific Aim 3: To conduct longitudinal analysis of the mechanisms of action of the integrated PN+SPI. To understand the mechanisms of change in the PN+SPI intervention, we will assess the theoretical purported targets (i.e., decreases in thwarted belongingness and increases in suicide-related coping skills). We hypothesize that participants assigned to the PN+SPI intervention will demonstrate clinically meaningful changes in the target variables relative to participants assigned to the SPI alone condition. Subsequently, these changes in proposed targets will predict changes in suicidal attempts.

ELIGIBILITY:
Inclusion Criteria:

1) age 15 to 29 years; 2) identifies as gay, lesbian, bisexual, transgender, genderqueer, asexual, pansexual, non-binary, or another non-exclusively heterosexual or cisgender identity, and/or reports same-gender romantic attraction, and/or reports same-gender sexual behavior in the past 12 months; 3) resides in Southern California; 4) speaks English; 5) is willing and able to provide informed consent; 6) reports suicidal ideation over the past two weeks, as indicated by the clinician-administered Columbia-Suicide Severity Rating Scale (C-SSRS) Baseline version; and 7) reports a lifetime history of one or more suicide attempts.

Exclusion Criteria:

1) Individuals with immediate intention to attempt suicide will be excluded.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Identify as gay, lesbian, bisexual, transgender, genderqueer, asexual, pansexual, non-binary, or another non-exclusively heterosexual or cisgender identity, and/or reports same-gender romantic attraction, and/or reports same-gender sexual behavior in the past 12 months.
Enrollment: 170 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | Presence or absence of suicide attempts in the full twelve-month following-up period
  Assess presence or absence of suicide attempts (i.e., actual, interrupted, or aborted) over the twelve-month follow-up period

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | Change from baseline suicidal ideation severity scores at 3 months, 6 months, and 12 months
  Assess suicidal ideation severity (5 items [yes/no]; scores range from 0 to 5 with higher scores indicating more severe suicidal ideation)
Columbia-Suicide Severity Rating Scale (C-SSRS) | Change from baseline suicidal ideation intensity scores at 3 months, 6 months, and 12 months
  Assess suicidal ideation intensity (5 items on 5-point scales; scores range from 0 to 25 with higher scores indicating more intense suicidal ideation)
The Interpersonal Needs Questionnaire-15 (INQ-15) - Thwarted Belongingness | Change from baseline thwarted belongingness scores at 3 months, 6 months, and 12 months
  Assess thwarted belongingness (9 items on 7-point scales; scores range from 9 to 63 with higher scores indicating greater thwarted belongingness)
Suicide-Related Coping Scale (SRCS) - Internal Coping Skills | Change from baseline suicide-related internal coping scores at 3 months, 6 months, and 12 months
  Assess suicide-related internal coping skills (7 items on 5-point scales; scores range from 0 to 28 with higher scores indicating better internal coping)
Suicide-Related Coping Scale (SRCS) - External Coping Skills | Change from baseline suicide-related external coping scores at 3 months, 6 months, and 12 months
  Assess suicide-related internal coping skills (7 items on 5-point scales; scores range from 0 to 28 with higher scores indicating better external coping)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Blashill, Ph.D., Principal Investigator — San Diego State University; Kristen J Wells, Ph.D., Principal Investigator — San Diego State University; Arjan van der Star, Ph.D., Study Director — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Background] Olfson M, Blanco C, Wall M, Liu SM, Saha TD, Pickering RP, Grant BF. National Trends in Suicide Attempts Among Adults in the United States. JAMA Psychiatry. 2017 Nov 1;74(11):1095-1103. doi: 10.1001/jamapsychiatry.2017.2582. PMID 28903161
- [Background] Ivey-Stephenson AZ, Crosby AE, Jack SPD, Haileyesus T, Kresnow-Sedacca MJ. Suicide Trends Among and Within Urbanization Levels by Sex, Race/Ethnicity, Age Group, and Mechanism of Death - United States, 2001-2015. MMWR Surveill Summ. 2017 Oct 6;66(18):1-16. doi: 10.15585/mmwr.ss6618a1. PMID 28981481
- [Background] Shepard DS, Gurewich D, Lwin AK, Reed GA Jr, Silverman MM. Suicide and Suicidal Attempts in the United States: Costs and Policy Implications. Suicide Life Threat Behav. 2016 Jun;46(3):352-62. doi: 10.1111/sltb.12225. Epub 2015 Oct 29. PMID 26511788
- [Background] Institute of Medicine (US) Committee on Lesbian, Gay, Bisexual, and Transgender Health Issues and Research Gaps and Opportunities. The Health of Lesbian, Gay, Bisexual, and Transgender People: Building a Foundation for Better Understanding. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK64806/ PMID 22013611
- [Background] Kann L, McManus T, Harris WA, Shanklin SL, Flint KH, Queen B, Lowry R, Chyen D, Whittle L, Thornton J, Lim C, Bradford D, Yamakawa Y, Leon M, Brener N, Ethier KA. Youth Risk Behavior Surveillance - United States, 2017. MMWR Surveill Summ. 2018 Jun 15;67(8):1-114. doi: 10.15585/mmwr.ss6708a1. PMID 29902162
- [Background] Miranda-Mendizabal A, Castellvi P, Pares-Badell O, Almenara J, Alonso I, Blasco MJ, Cebria A, Gabilondo A, Gili M, Lagares C, Piqueras JA, Roca M, Rodriguez-Marin J, Rodriguez-Jimenez T, Soto-Sanz V, Vilagut G, Alonso J. Sexual orientation and suicidal behaviour in adolescents and young adults: systematic review and meta-analysis. Br J Psychiatry. 2017 Aug;211(2):77-87. doi: 10.1192/bjp.bp.116.196345. Epub 2017 Mar 2. PMID 28254960
- [Background] Stanley B, Brown GK, Brenner LA, Galfalvy HC, Currier GW, Knox KL, Chaudhury SR, Bush AL, Green KL. Comparison of the Safety Planning Intervention With Follow-up vs Usual Care of Suicidal Patients Treated in the Emergency Department. JAMA Psychiatry. 2018 Sep 1;75(9):894-900. doi: 10.1001/jamapsychiatry.2018.1776. PMID 29998307
- [Background] Labouliere CD, Stanley B, Lake AM, Gould MS. Safety Planning on Crisis Lines: Feasibility, Acceptability, and Perceived Helpfulness of a Brief Intervention to Mitigate Future Suicide Risk. Suicide Life Threat Behav. 2020 Feb;50(1):29-41. doi: 10.1111/sltb.12554. Epub 2019 May 21. PMID 31112330
- [Background] Cramer RJ, Kapusta ND. A Social-Ecological Framework of Theory, Assessment, and Prevention of Suicide. Front Psychol. 2017 Oct 9;8:1756. doi: 10.3389/fpsyg.2017.01756. eCollection 2017. PMID 29062296
- See also: 10 Leading Causes of Death, United States: 2016, All Races, Both Sexes — https://www.cdc.gov/nchs/products/databriefs/db293.htm
- See also: Safety Planning Intervention: A Brief Intervention to Mitigate Suicide Risk — https://doi.org/10.1016/j.cbpra.2011.01.001